CLINICAL TRIAL: NCT00917748
Title: A Prospective, Randomised, Double-Blind, Placebo-Controlled Phase III Study of Modafinil to Improve Fatigue and Quality of Life in Patients Treated With Docetaxel-Based Chemotherapy for Metastatic Breast or Prostate Cancer
Brief Title: Study With Modafinil in Patients Treated With Docetaxel-Based Chemotherapy for Metastatic Breast or Prostate Cancer (MOTIF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOCET_L_04203
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Prostatic Neoplasms; Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): docetaxel chemotherapy + modafinil 100 mg capsules
  Interventions: Drug: DOCETAXEL(XRP6976) + MODAFINIL; Drug: Modafinil
- 2 (Placebo Comparator): docetaxel chemotherapy + placebo (lactose) capsules (matched to modafinil drug)
  Interventions: Drug: DOCETAXEL(XRP6976) + MODAFINIL; Drug: Placebo of Modafinil

INTERVENTIONS:
Drug: DOCETAXEL(XRP6976) + MODAFINIL — arm 1: best supportive care (docetaxel chemotherapy) plus modafinil 200mg mane daily arm 2: best supportive care (docetaxel chemotherapy) plus placebo of modafinil 200mg mane daily
Drug: Modafinil — best supportive care (docetaxel chemotherapy) plus modafinil 200mg mane daily
  Arms: 1
Drug: Placebo of Modafinil — Best supportive care (docetaxel chemotherapy) + placebo capsules one daily-mane (before noon)
  Arms: 2

SUMMARY:
The primary objective is:

* To determine the efficacy of modafinil in the reduction of fatigue in patients with metastatic breast or prostate cancer undergoing docetaxel-based chemotherapy

The secondary objectives are:

* To determine the effect of modafinil on quality of life (QoL) during docetaxel-based chemotherapy
* To determine the effect of modafinil on patients physical activity level, functional status, number of chemotherapy cycles tolerated, sleep disturbance and depression, during docetaxel-based chemotherapy
* To investigate the impact of tumour type, patient physical activity level, functional status, sleep disturbance and depression on the efficacy of modafinil at improving fatigue and quality of life during docetaxel-based chemotherapy.
* To determine the safety and tolerability of modafinil during docetaxel-based chemotherapy

ELIGIBILITY:
Inclusion criteria:

* Treatment with q3w (every three weeks) docetaxel-based chemotherapy for metastatic breast or prostate cancer at a minimum dose of 50 mg/m2
* Completed at least two cycles of chemotherapy and intention to treat the patient with at least two further cycles of docetaxel-based chemotherapy
* Fatigue > or = to 4 on the MD Anderson Symptom Inventory fatigue assessment scale during the previous docetaxel chemotherapy cycle
* SPHERE somatic (SOMA) subscale score > or = to 3
* Worsening of fatigue after commencement of docetaxel chemotherapy
* Haemoglobin (Hb)> or = to 10 g/dL within two weeks before randomisation

Exclusion criteria:

* Unable to complete the MD Anderson Symptom Inventory fatigue assessment scale or Functional Assessment of Chronic Illness Therapy-Fatigue Quality of Life survey
* Require docetaxel chemotherapy dose reduction to less than 50 mg/m2
* History of chronic fatigue condition
* Uncontrolled hypertension (blood pressure > or = to 150/90 mm Hg
* Known hypersensitivity / intolerance to modafinil or any of the excipients
* Pregnant women
* Psychological, familial, sociological, or geographical conditions that do not permit treatment or medical follow-up and / or prohibit compliance with the study protocol
* Any serious concomitant illness that, in the opinion of the Investigator, would preclude a patient from participating in the study
* Non-English speaking

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Fatigue scores daily assessed using the 11-point (0-10) 0 is the lower score and 10 is the highest. this score is calculated using the MD Anderson Symptom Inventory | From baseline to the end of study (week 12)

SECONDARY OUTCOMES:
Patient quality of life weekly assessed by using the self-administered Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Quality Of Life survey | From baseline to the end of study (week 12)
Fatigue assessed by using the self-administered six-item somatic subscale (SOMA) of the Somatic and Psychological Health Report (SPHERE) questionnaire | At screening and from visit 6 (week 3) of treatment to end of study (week 12)
Sleep quality assessed by using the self-administered Pittsburgh Sleep Quality Index (PSQI) questionnaire | At baseline and from visit 6 (week 3) to end of study (week 12)
Functional status will be determined using the self-administered Medical Outcomes Study - Short Form Health Survey (SF-36) | At baseline and from visit 6 (week 3) to end of study (week 12)
Depression assessed using seven depression-related questions from the self-administered Hospital Anxiety and Depression (HAD) assessment subscale. Patient with depression will be defined as having the HAD-D> or = 8 | At baseline and last visit= end of study (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna DUFFY, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia

REFERENCES:
- [Derived] Hovey E, de Souza P, Marx G, Parente P, Rapke T, Hill A, Bonaventura A, Michele A, Craft P, Abdi E, Lloyd A; MOTIF investigators. Phase III, randomized, double-blind, placebo-controlled study of modafinil for fatigue in patients treated with docetaxel-based chemotherapy. Support Care Cancer. 2014 May;22(5):1233-42. doi: 10.1007/s00520-013-2076-0. Epub 2013 Dec 17. PMID 24337761